CLINICAL TRIAL: NCT00786565
Title: Clinical Evaluation of a New Aspheric Intraocular Lens. A Prospective, Multi-Center, Comparative Study.
Brief Title: Clinical Evaluation of a New Aspheric Intraocular Lens.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 001/04
Record Dates: First submitted 2008-11-03; First posted 2008-11-06 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advanced Akreos Adapt (Experimental): Advanced Akreos Adapt Aspheric Intraocular Lens (IOL).
  Interventions: Device: Advanced Akreos Adapt in one operated eye.
- Akreos Adapt (Experimental): Akreos Adapt Spherical Intraocular Lens (IOL).
  Interventions: Device: Akreos Adapt in fellow operated eye.

INTERVENTIONS:
Device: Advanced Akreos Adapt in one operated eye. — Cataract surgery to implant the assigned IOL according to randomized schedule.
  Arms: Advanced Akreos Adapt
Device: Akreos Adapt in fellow operated eye. — Cataract surgery to implant the assigned IOL according to randomized schedule.
  Arms: Akreos Adapt

SUMMARY:
This study evaluates the visual performance and occurrence of posterior capsular opacification after implantation of a new aspherical intraocular lens compared with a control spherical lens of otherwise identical design.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinically documented diagnosis of bilateral cataract (either cortical, nuclear, subcapsular or a combination) liable to benefit from standard cataract surgery.
* Patients must be undergoing primary cataract surgery with IOL in-the-bag implantation, requiring a IOL power from 10 to 30 diopters.

Exclusion Criteria:

* Patients with corneal damage.
* Patients with any anterior segment pathology for which extracapsular phacoemulsification cataract surgery would be contraindicated.
* Patients with any ocular pathology, other than the cataract, having repercussions on visual function:

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 12/15/2004 and ended on 04/28/2006. This study was conducted at 5 European sites.
Pre-assignment Details: Planned enrollment was to consist of 120 subjects, due to difficulties in enrolling subjects within the designated 6 month enrollment window 75 subjects were entered into the study for a total of 150 treated eyes.
Groups:
- Akreos Intraocular Lens: Subjects randomised to receive Akreos Advanced Optic Aspheric Intraocular Lens in one eye and Akreos Adapt Spherical Intraocular Lens in the fellow eye.
Period: Enrollment Prior to Surgery
Arm/Group | Akreos Intraocular Lens
Started | 75
Completed | 69 (69 participants - Akreos Advanced Optic Lens in one eye and Akreos Adapt Lens in the fellow eye.)
Not Completed | 6
Not completed — Site Closed | 3
Not completed — Protocol Violation | 3
Period: Post Surgery
Arm/Group | Akreos Intraocular Lens
Started | 69
Completed | 67 (67 Participants (134 eyes) completed the study.)
Not Completed | 2
Not completed — Abnormal macular pucker | 1
Not completed — Adapt AO implanted posterior side up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Akreos Intraocular Lens
Number analyzed (Participants) | 69
Age, Customized [Mean (Standard Deviation); unit: years] — 69 participants (138 eyes)were randomised to receive Akreos Advanced Optic Aspheric Intraocular Lens in one eye (69 eyes) and Akreos Adapt Spherical Intraocular Lens in the fellow eye (69 eyes).
  years
    Between 50 and 85 years | 73.0 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 32
Region of Enrollment [Number; unit: participants]
  Europe | 69

OUTCOME MEASURES:

1. Primary Outcome: Low Contrast Best Corrected Visual Acuity Following Cataract Surgery
Description: Low contrast best corrected visual acuity (ability to distinguish objects on a similarly colored or shaded background) 3 months following cataract surgery.
Time Frame: 3 months
Population: Number of participants 67 total with 67 eyes in each group, full analysis set, all randomized participants who had cataract surgery one intraocular lens (IOL) in each eye, and who had at least one baseline value and one post-baseline value for efficacy.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Akreos Advanced Optics: Akreos Advanced Optics Intraocular Lens
- Akreos Adapt: Akreos Adapt Intraocular Lens
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 67 | 67
LogMAR | 0.22 (0.096) | 0.24 (0.131)

2. Primary Outcome: Low Contrast Uncorrected Visual Acuity Following Cataract Surgery
Description: Low contrast uncorrected visual acuity 3 months post cataract surgery
Time Frame: 3 months
Population: Full analysis set, all randomized participants who had cataract surgery one intraocular lens (IOL) in each eye, and who had at least one baseline value and one post-baseline value for efficacy
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 68 | 68
LogMAR | 0.33 (0.163) | 0.35 (0.191)

3. Primary Outcome: Photopic Contrast Sensitivity
Description: The mean photopic (day light) contrast sensitivity for each spatial frequency (cycle per degree-CPD) (1.5, 3.0, 6.0, 12.0 and 18 cpd)
Time Frame: 3 months
Population: All patients who had cataract surgery and who have at least one baseline value and one post-baseline value for efficacy criteria.
Measure: Mean (Standard Deviation); unit: Log 10
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 68 | 68
Log 10
  Photopic Contrast Sensitivity - 1.5 | 44.4 (22.5) | 41.1 (21.3)
  Photopic Contrast Sensitivity - 3.0 | 78.3 (36.2) | 81.1 (38.5)
  Photopic Contrast Sensitivity - 6.0 | 89.6 (48.4) | 86.4 (45.5)
  Photopic Contrast Sensitivity - 12.0 | 29.3 (18.3) | 26.7 (20.4)
  Photopic Contrast Sensitivity - 18.0 | 11.4 (9.6) | 10.1 (10.7)

4. Secondary Outcome: High Contrast Visual Acuity
Description: High contrast visual acuity (ability to distinguish objects of contrasting color such as black on white) uncorrected and best corrected visual acuity.
Time Frame: 1 month
Population: Patients without missing values for HCVA logmar at pre-operative and post operative at 1 month control.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 66 | 66
LogMAR
  Uncorrected | 0.13 (0.20) | 0.18 (0.21)
  Best Corrected | 0.02 (0.13) | 0.05 (0.14)

5. Secondary Outcome: High Contrast Visual Acuity Uncorrected
Time Frame: 3 months
Population: Patients without missing values for UHCVA logmar at pre-operative and post operative at 1 month control.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 66 | 67
LogMAR | 0.15 (0.19) | 0.18 (0.22)

6. Secondary Outcome: High Contrast Visual Acuity Best Corrected
Time Frame: 3 months
Population: Patients without missing values for BHCVA logmar at pre-operative and post operative at 1 month control.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 64 | 66
LogMAR | 0.03 (0.12) | 0.04 (0.13)

7. Secondary Outcome: High Contrast Visual Acuity
Time Frame: 12 months
Population: Patients without missing values for HCVA logmar at pre-operative and post operative at 1 month control.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 60 | 60
LogMAR
  Uncorrected | 0.17 (0.19) | 0.22 (0.22)
  Best Corrected | 0.05 (0.13) | 0.07 (0.13)

8. Primary Outcome: Mesoptic Contrast Sensitivity
Description: The mean mesoptic (low light) contrast sensitivity for each spatial frequency (cycle per degree-CPD) (1.5, 3.0, 6.0, 12.0 and 18 cpd)
Time Frame: 3 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 68 | 67
Log 10
  Mesopic Contrast Sensitivity - 1.5 | 51.2 (27.0) | 47.4 (25.4)
  Mesopic Contrast Sensitivity - 3.0 | 65.6 (35.6) | 58.1 (35.0)
  Mesopic Contrast Sensitivity - 6.0 | 52.9 (33.5) | 45.6 (29.4)
  Mesopic Contrast Sensitivity - 12.0 | 9.5 (10.2) | 9.5 (13.0)
  Mesopic Contrast Sensitivity - 18.0 | 2.7 (4.9) | 2.0 (3.3)

9. Primary Outcome: Posterior Capsule Opacification Score
Description: Posterior Capsule Opacification Score (PCO), Density of opacification measured from 0-4 (1=minimal and 4=severe) and area of opacification measured from 0-1 (0=no opacification and 1=posterior capsule opacification required a treatment). Results (EPCO) were computer calculated by multiplying density by area of opacification.
Time Frame: 24 months
Population: The EPCO score, evaluated by an independent observer using retro-illumination pictures, all pictures available. Measured in a 3mm and 6mm optic area.
Measure: Mean (Standard Deviation); unit: EPCO Score
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 34 | 30
EPCO Score
  PCO Score 3mm | 0.05 (0.14) | 0.14 (0.24)
  PCO Score 6mm | 0.12 (0.24) | 0.20 (0.31)

10. Secondary Outcome: High Contrast Visual Acuity Uncorrected
Time Frame: 24 Months
Population: Patients without missing values for UHCVA logmar at pre-operative and post operative at 1 month control.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 55 | 55
LogMar | 0.22 (0.18) | 0.27 (0.23)

11. Secondary Outcome: High Contrast Visual Acuity Best Corrected
Time Frame: 24 Months
Population: Patients without missing values for best corrected HCVA logmar at pre-operative and post operative at 1 month control.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 52 | 52
LogMar | 0.11 (0.14) | 0.15 (0.19)

12. Secondary Outcome: Low Contrast Visual Acuity
Description: Uncorrected Low contrast visual acuity - LogMar visual acuity value
Time Frame: 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 68 | 68
LogMar
  Uncorrected | 0.33 (0.17) | 0.36 (0.19)
  Best Corrected | 0.21 (0.13) | 0.24 (0.12)

13. Secondary Outcome: Contrast Sensitivity Photopic 1.5cpd
Description: The mean photopic (day light) contrast sensitivity were to be compared between both IOLs for each special frequency (1.5, 3.0, 6.0, 12.0 and 18 cpd)
Time Frame: 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 67 | 67
Log 10 | 39.2 (20.80) | 39.9 (20.08)

14. Secondary Outcome: Contrast Sensitivity Photopic
Description: as for outcome 13
Time Frame: 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 66 | 66
Log 10
  Photopic contrast sensitivity - 3.0 | 76.6 (36.38) | 64.0 (27.83)
  Photopic contrast sensitivity - 6.0 | 92.4 (46.34) | 70.5 (39.15)
  Photopic contrast sensitivity - 12.0 | 30.3 (21.46) | 22.3 (17.60)
  Photopic contrast sensitivity - 18.0 | 11.0 (9.12) | 8.3 (8.90)

15. Secondary Outcome: Contrast Sensitivity Mesoptic 1.5 Cpd
Description: The mean mesopic (dim light) contrast sensitivity were to be compared between both IOLs for each special frequency (1.5, 3.0, 6.0, 12.0 and 18 cpd)
Time Frame: 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 67 | 67
Log 10 | 46.6 (25.21) | 40.8 (21.74)

16. Secondary Outcome: Contrast Sensitivity Mesoptic
Description: as for outcome 15
Time Frame: 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 66 | 66
Log 10
  Mesoptic contrast sensitivity - 3.0 | 58.2 (28.08) | 51.5 (29.57)
  Mesoptic contrast sensitivity - 6.0 | 55.9 (40.56) | 39.4 (28.32)
  Mesoptic contrast sensitivity - 12.0 | 9.2 (10.29) | 6.7 (10.21)
  Mesoptic contrast sensitivity - 18.0 | 2.8 (4.97) | 2.2 (3.84)

17. Secondary Outcome: Posterior Capsule Opacification
Description: as for outcome 9
Time Frame: 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: EPCO Score
Arm/Group | Akreos Advanced Optics | Akreos Adapt
Number analyzed (Participants) | 40 | 39
EPCO Score
  PCO Score - 3mm | 0.03 (0.095) | 0.06 (0.133)
  PCO Score - 6 mm | 0.07 (0.148) | 0.13 (0.195)

ADVERSE EVENTS:
Time Frame: Ocular adverse events were measured over 24 month study period.
Groups:
- Akreos Advanced Intraocular Lenses; Akreos Adapt Intraocular Lens: Akreos Advanced Optic Aspheric Intraocular Lens in one eye and Akreos Adapt Spherical Intraocular Lens in the fellow eye.
Arm/Group | Akreos Advanced Intraocular Lenses | Akreos Adapt Intraocular Lens
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less